CLINICAL TRIAL: NCT05318235
Title: Virus Interactions in the Respiratory Tract; a Cohort Study With Children
Acronym: VIOOL
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Patricia Bruijning-Verhagen, Principal investigator, UMC Utrecht
Other Study IDs: NL78424.041.21
Record Dates: First submitted 2022-03-17; First posted 2022-04-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Tract Infections; Coinfection
Keywords: Child; Viral interference
MeSH Terms: conditions — Respiratory Tract Infections; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Midturbinate nasal swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children: Children between 6 weeks and 4 years of age who have a older sibling or attend day care
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Rationale: Prevention of virus induced acute respiratory infection (ARI) is a public health priority. As different respiratory virus infections can interact with each other, occurrence of one virus may influence occurrence of other virus infections. Such interactions can have implications for the effects of vaccination on non-target diseases. In this project, we will quantify such interactions between respiratory viruses by longitudinally studying a cohort of young children.

Objective: To quantify the strength and direction of interactions between important respiratory virus infections in young children.

Study design: This is a prospective observational cohort study.

Study population: Children between 6 weeks and 4 years of age residing in the Utrecht area of the Netherlands.

Main study parameters/endpoints: Frequency, timing and sequences of occurrence of respiratory virus infections will be studied for each participant using weekly collected nasal specimens during 16 weeks follow-up. Detection will be based on PCR testing for a panel of common respiratory viruses. From these data, estimation of virus interaction parameters will be based on self-controlled-case series analysis.

Nature and extend of the burden and risks associated with participation, benefit and group relatedness: This study is observational in nature. There will be no direct benefit to research participants. The study includes biological sampling. The results of the tests done on these samples may not contribute to improving the participant's health. Minimal inconvenience and discomfort to the participant may arise from study visits and biological sampling.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 weeks and 4 years AND
* 1) have older siblings or 2) attend daycare. AND
* Live within 30 minutes drive from UMCU (by car), have access to a fever thermometer and a freezer were biological samples can be temporarily stored

Exclusion Criteria:

* recurrent respiratory tract infections and are treated with antibiotic prophylaxis OR
* known immunodeficiency OR
* chronic lung disease that increases susceptibility to infection (e.g. cystic fibrosis) OR
* congenital anomalies of the airways
* Parents/guardians have insufficient comprehension of Dutch language (all study communication and questionnaires are in Dutch language)

Ages: 6 Weeks to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample of children living within the region of Utrecht.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Strength of viral interactions | Samples and data collected during 16 weeks of follow-up
  To quantify the strength of interactions between common respiratory virus infections in young children.
Direction of viral interactions | Samples and data collected during 16 weeks of follow-up
  To quantify the direction of interactions between common respiratory virus

SECONDARY OUTCOMES:
To quantify relative change in disease severity due to viral interactions. | Samples and data collected during 16 weeks of follow-up
  This will be measured as changes in disease severity scores of one virus infection upon recent exposure to another virus infection
To estimate the seasonal incidence rates of both symptomatic and asymptomatic infection by common respiratory viruses in young children | Samples and data collected during 16 weeks of follow-up
To estimate the probability of symptomatic versus asymptomatic infection per respiratory virus and host factors influencing this. | Samples and data collected during 16 weeks of follow-up
To quantify the changes in viral exposure in the pandemic-to-post-pandemic transition period and study effects of these changes on viral interaction patterns | Samples and data collected during 16 weeks of follow-up

OTHER OUTCOMES:
To explore local inflammatory responses that could mediate observed virus interaction patterns and effects on disease severity | Samples and data collected during 16 weeks of follow-up
To explore the nasal microbiological community in young children | Samples and data collected during 16 weeks of follow-up
To examine immunity against respiratory viruses in saliva | Samples and data collected during 16 weeks of follow-up
To explore viral-bacterial interactions in young children | Samples and data collected during 16 weeks of follow-up
To study the effect of pandemic exposure on respiratory infections and local inflammatory responses | Samples and data collected during 16 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bruijning, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided